CLINICAL TRIAL: NCT01363778
Title: A Phase 1, Open-label Study to Evaluate The Effect of Ketoconazole on the Pharmacokinetics, Safety, and Tolerability of a Single Dose of Tivozanib in Healthy Subjects
Brief Title: A Phase 1 Study to Evaluate The Effect of Ketoconazole on the Pharmacokinetics of Tivozanib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-11-116
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: AV-951; Tivozanib; Healthy Subjects; ketoconazole; Pharmacokinetics
MeSH Terms: interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tivozanib (Experimental): Tivozanib is a novel and potent pan-vascular endothelial growth factor (VEGF) receptor (VEGFR) tyrosine kinase inhibitor with potent activity against all 3 VEGFRs (VEGFR-1, -2, and -3). In nonclinical models and studies performed in humans, tivozanib has shown strong antiangiogenesis and antitumor activity.
  Interventions: Drug: tivozanib

INTERVENTIONS:
Drug: tivozanib — Tivozanib is a novel and potent pan-vascular endothelial growth factor (VEGF) receptor (VEGFR) tyrosine kinase inhibitor with potent activity against all 3 VEGFRs (VEGFR-1, -2, and -3). In nonclinical models and studies performed in humans, tivozanib has shown strong antiangiogenesis and antitumor activity.

SUMMARY:
This study is designed to evaluate the effect ketoconazole on the Pharmacokinetic profile of tivozanib.

DETAILED DESCRIPTION:
This Phase 1, open-label, two-period, single-sequence study is designed to evaluate the effect of steady-state ketoconazole on the PK profile, safety, and tolerability of a single 1.5-mg tivozanib dose. On Day 1 of the first period, subjects will receive a single 1.5-mg dose of tivozanib and remain at the unit for at least 48 hours postdose followed by outpatient visits for PK sampling and safety assessments up to 3 weeks postdose. For Period 2, subjects will be administered 400 mg of ketoconazole once daily (QD) for 3 days. On the 4th day of Period 2, 1.5mg of tivozanib will be administered with 400mg of ketoconazole. PK sampling will continue for 3-weeks postdose while the subjects continue to receive 400mg of ketoconazole daily. An end of study visit will be completed 1-week after the last dose of ketoconazole.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, between 18 and 55 years of age, inclusive.
2. Body mass index (BMI) within the range of 18.5 to 31.0 kg/m2, inclusive.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs.
4. Clinical laboratory evaluations (including a chemistry panel comprised of 20 analytes [Chem-20, includes liver function tests; fasted approximately 10 hours], complete blood count [CBC], and urinalysis) not exceeding 2 x upper limit of normal (ULN) or < lower limit of normal (LLN), unless deemed not clinically significant by the Investigator.
5. Nonsmokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to Screening), verified by a cotinine test at Screening and each study period Check-in.
6. Negative test for selected drugs of abuse at Screening (does not include alcohol) and at each study period Check-in (does include alcohol; Appendix A).
7. Negative hepatitis panel (including hepatitis B virus surface antigen [HBsAg] and hepatitis C virus antibody [anti-HCV] and negative human immunodeficiency virus [HIV] antibody screens; Appendix A).
8. Females who are not pregnant, non-lactating, and either postmenopausal for at least 1 year, surgically sterile (eg, tubal ligation, hysterectomy) for at least 90 days prior to Screening, or agree to use at least 1 of the following forms of contraception from informed consent until 45 days after Study Completion: a non-hormonal intrauterine device with spermicide; female condom with spermicide; contraceptive sponge with spermicide; diaphragm with spermicide; cervical cap with spermicide; a male sexual partner who agrees to use a male condom with spermicide; or a sterile sexual partner. For all females, a serum pregnancy test result must be negative at Screening and at each study period Check-in.
9. Male subjects who are either sterile or agree to use, during the period from informed consent until 45 days following Study Completion, 1 of the following approved methods of contraception: a double barrier method (eg, male condom with spermicide, use by female sexual partner of an intrauterine device with spermicide, a female condom with spermicide, contraceptive sponge with spermicide, a diaphragm with spermicide, or use of a cervical cap with spermicide); a sterile sexual partner; a female sexual partner using an intravaginal system (eg, NuvaRing®); or a partner using an oral, implantable, transdermal, or injectable contraceptives.
10. Able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

1. Significant history or clinical manifestation of any significant metabolic/endocrine, allergic, dermatological, hepatic, renal, hematological, pulmonary, immune, cardiovascular, gastrointestinal, genitourinary, neurological, or psychiatric disorder (as determined by the Investigator or Sponsor's Medical Monitor).
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
3. History of stomach or intestinal surgery, nephrectomy, cholecystectomy, or resection that would potentially alter absorption and/or excretion of orally administered drugs as determined by the Investigator (appendectomy and/or hernia repair may be allowed).
4. Diagnosis of alcoholism or drug addiction within 1 year prior to Period 1 Check-in.
5. Participation in any other investigational drug study in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer, prior to Period 1 Check-in.
6. Use of any prescription medications or products within 14 days prior to Period 1 Check-in.
7. Use of any over-the-counter (OTC), non-prescription, systemic preparations (including vitamins, minerals, and phytotherapeutic, herbal, dietary supplements, or plant derived preparations) within 7 days prior to each study period Check-in.
8. Consumption of food or beverages containing alcohol, grapefruit, Seville orange, or caffeine within 72 hours prior to each study period Check-in.
9. Use of known hepatic or renal clearance altering agents (eg, ketoconazole, erythromycin, cimetidine, barbiturates, phenothiazines, or herbal/plant derived preparations such as St. John's Wort) for a period of 60 days prior to Period 1 Check-in.
10. Poor peripheral venous access.
11. Donation of blood ≥ 250 mL from 30 days prior to Period 1 Check-in until Study Completion, inclusive, or of plasma from 2 weeks prior to Period 1 Check-in until Study Completion, inclusive.
12. Receipt of blood products within 2 months prior to Period 1 Check-in.
13. Blood pressure greater than 140/90 mmHg confirmed by repeat at Screening or at Period 1 Check-in. Up to 2 repeats may be conducted.
14. History of azole antifungal hypersensitivity.
15. Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To examine the effect of steady-state ketoconazole on the pharmacokinetics (PK) of a single dose of 1.5 mg of tivozanib in healthy subjects. | Planned Enrollment/Screening Duration: Approximately 4 weeks.
  Blood samples for PK analysis of serum tivozanib levels will be collected for a 3-week period following each dose.
To assess the safety and tolerability of tivozanib administered alone and in the presence of steady-state ketoconazole in healthy subjects. | Planned Enrollment/Screening Duration: Approximately 4 weeks.
  Safety assessments will be completed by evaluation of physical exam, ECGs, laboratory assessments and adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States